CLINICAL TRIAL: NCT07293507
Title: Effects of Modified Otago Exercises Versus Neuromuscular Dynamic Stabilization Exercises on Balance and Activities of Daily Living in Patients With Diabetic Peripheral Neuropathy
Brief Title: MOE and DNSE Effects on Balance and Activities of Daily Living Diabetic Peripheral Neuropathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7424 ZUNAIRA SALEEM BUTT
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Diabetes Mellitus Diabetic Peripheral Neuropathy Modified Otago Exercise Dynamic Neuromuscular Stabilization Berg Balance Scale Balance Training.
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Modified Otago Exercises
  Interventions: Other: Modified Otago Exercises
- Group B (Experimental): Dynamic Neuromuscular Stabilization Exercises
  Interventions: Other: Dynamic neuromuscular stabilization exercises

INTERVENTIONS:
Other: Modified Otago Exercises — The 30-minute Otago Exercise Program, involving both balance and strength training, followed by further 15 minutes of walking as part of the modified-OEP group intervention will be given. The 15-minute walk will be completed by walking continuously at an appropriate pace in the approximately 15-meter exercise room. Participants will be told to walk 15 meters, execute a U-turn to the left, walk 15 meters, and then execute a U-turn to the right at the next turning point to create the same effect on the stated benefit of symmetry while turning left and right. For twelve weeks, the intervention will be given three times a week.
  Arms: Group A
Other: Dynamic neuromuscular stabilization exercises — The Dynamic neuromuscular stabilization exercises (DNS) twice a week for 60 minutes each time for 12 weeks. A five-minute warm-up, a fifty-minute exercise plan, and a five-minute cool-down comprised the program. Static stretching was used for the cool-down and dynamic stretching for the warm-up. DNS training is conducted in three levels. Level 1 (1 to 4 weeks) includes: (1) dynamic stretching (2) baby rock (3) breathing (4) rolling. Level 2 (5 to 8 weeks) includes: (1) oblique sit (2) aqua bag tripod (3) aqua bag sitting (4) aqua bag kneeling. Level 3 (9 to 12 weeks) include: (1) aqua bag high kneeling (2) static stretching (3) aqua bag standing
  Arms: Group B

SUMMARY:
The purpose of this study is to compare the impact of Modified Otago Exercises and Dynamic Neuromuscular Stabilization Exercises on patients with diabetic peripheral neuropathy (DPN) using valid tools such as the Berg Balance Scale and the Katz Index of Independence in ADL. The results of our study will be helpful for clinical decision-making in terms of selecting specific physiotherapy treatment techniques in an attempt to improve their function, reduce their falls, and improve their independence specific to diabetes neuropathy.

DETAILED DESCRIPTION:
Research into therapeutic exercise for patients with diabetic peripheral neuropathy (DPN) has grown over the past decade due to the increasing recognition of non-pharmacological strategies for reducing fall risk and restoring function. DPN is associated with altered gait, diminished proprioception, and increased postural sway, making balance-specific exercise programs a critical area of intervention.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age and elderly.
* The Timed Up and Go score exceeds 10 seconds.
* Both men and women
* Individuals with type 2 diabetes and DPN.
* Patients diagnosed with diabetes from last 5 Years.
* Patients diagnosed with diabetic peripheral neuropathy with scores ≥ 4 on Michigan Neuropathy Screening Instrument (MNSI)
* Individuals with an ability to walk independently.

Exclusion Criteria:

* Individuals with neuropathies that are not caused by diabetes.
* Individuals with any neurological disorders that may affect their ability to balance.
* Participants suffering from any musculoskeletal disorders that result in discomfort and instability.
* A history of acute and chronic physiological, psychological, and mental disorders that may prevent exercise.
* Participants with unrelated orthopedics, surgical, or health conditions that impair physical movement and equilibrium, such as severe diabetic retinopathy were eliminated, as were those with active foot issues.
* Patients having serious complications of diabetes, such as amputation and patients who are unable to complete the entire program.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 36 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Katz Index of Independence in Activities of Daily Living | Baseline, after 6th week, after 12th week
  The Katz Index of Independence in Activities of Daily Living (ADL) is a tool that assesses a person's ability to perform six basic self-care tasks: bathing, dressing, toileting, transferring, continence, and feeding
Berg Balance Scale | Baseline, After 6th week, After 12th week
  The Berg Balance Scale (BBS) is a 14-item test that assesses an individual's static and dynamic balance through a series of tasks, such as sitting to standing, reaching, and turning.

CONTACTS AND LOCATIONS:
Overall Officials: Sana Riaz, Nmpt, Principal Investigator
Locations (1):
- imran idrees teaching hospital daska Road sialkot, Dar ul shifa hospital sialkot, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No